CLINICAL TRIAL: NCT05872581
Title: The Effectiveness of a Multicomponent Education Program of Hand Hygiene in Nursing Students: a Randomized Controlled Trial
Brief Title: Education Program of Hand Hygiene for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr YANG Lin, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSEARS20230103002
Record Dates: First submitted 2023-04-25; First posted 2023-05-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hand Hygiene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hand scanner instant feedback (Experimental): Hand scanner results only but no training videos will be provided.
  Interventions: Behavioral: Hand scanner instant feedback
- Video training (Experimental): A training video only but no hand scanner results will be provided.
  Interventions: Behavioral: Video training
- Hand scanner and Video training (Experimental): Both hand scanner results and a training video will be provided.
  Interventions: Behavioral: Hand scanner instant feedback; Behavioral: Video training
- Control group without intervention (No Intervention): No hand scanner results or training videos will be provided.

INTERVENTIONS:
Behavioral: Hand scanner instant feedback — Participants will be informed about their hand scanner results of the first hand washing attempt to get individualized feedback about their hand wash performance.
  Arms: Hand scanner and Video training; Hand scanner instant feedback
Behavioral: Video training — Participants will watch a training video about the 7 steps of hand washing after the first hand washing attempt.
  Arms: Hand scanner and Video training; Video training

SUMMARY:
The goal of this observational study is to design and test a multicomponent education program of hand hygiene in nursing students. The main aims are:

1. conduct a randomized controlled trial (RCT) to test the effectiveness of this program on knowledge and practice of hand hygiene in nursing students;
2. evaluate the effects of each component and collect feedbacks from participants.

Participants will be randomly assigned into the three intervention: Group A (Hand scanner instant feedback) , Group B (Video training), Group C (Hand scanner + Video training) , and Group D (Control group without intervention). Pre- and post-intervention assessment will be used to evaluate the effectiveness of the program and individual components.

DETAILED DESCRIPTION:
Background

The ongoing COVID-19 pandemic has posed serious threats to public health worldwide. Although children have mild symptoms, they have been found to more likely transmit the virus within the household than the other age groups. The importance of hand hygiene cannot be underestimated in both healthcare and community settings. The promotion of hand hygiene is the best practices in preventing health care-associated infection. It has been estimated that hand hygiene could reduce over 500000 attributable deaths per year. It was found that the annual economic impact of health care-associated infection in the US was approximately US$6.5 billion in 2004 and every US$1 spent on hand hygiene promotion could result in a US$23.7 benefit. Education plays a key role in setting a good practice base in hand hygiene.

The traditional training methods for nursing students include in-class lecture and practical, but students seldom receive individualized instructions and feedbacks due to limited manpower and facilities. Hence, there is an urgent need of designing an automated and individualized education program. This study aims to design and test a multicomponent education program of hand hygiene in nursing students. Specifically, this program has two components: 1) training videos according to the WHO guidelines on hand hygiene in health care; 2) a hand scanner used for students to immediately visualize the missing spots of hand hygiene.

If demonstrated effective, this program can be integrated into the curriculum of nursing students as an e-learning approach. In future, this system can also be used at point-of-care for real-time monitoring and audit of healthcare workers in other healthcare settings.

Subject recruitment

The investigators will recruit all year one nursing students from the Bachelor of Nursing and Bachelor of Mental Health Nursing program in School of Nursing (total number is approximately 320). The participants will subscribe a timeslot of training sessions. All participants who attend the same session will be assigned to the same group by cluster randomization. A statistician will assign the groups in advance by a random number generator. The participants will not be informed about their group before arriving the study site.

The investigators calculated the statistical power for cluster randomized controlled trial. Since the total number is fixed to 320 and each cluster has 4 participants, there will be a total of 80 clusters which are equally divided into four groups. It is assumed that the standard deviation of subjects is 2.00, the intracluster correlation coefficient is 0.010, and the coefficient of variation of cluster sizes is 0.500. The sample size of 320 can achieve 87% power to detect a difference between the group means of at least 1 in a two-sided t-test with a significance level of 0.050.

Pre-intervention assessment

During the site visit, the participants will sign a consent form first and be asked to fill in a questionnaire on knowledge and practice of hand hygiene.

Participants will need to put fluorescent powder on both of their hands and then perform hand washing using liquid soap without any instructions (1st hand washing attempt). The camera installed above the hand-wash basins will take videos of both hands (no face nor other parts of the body) during this procedure. After washing hands, participants will need to scan fluorescent powder remained on their hands in a hand scanner (The Semmelweis Scanner™). The recorded hand washing videos will be used to train the AI algorithms for automatic image processing and assessments. Two IPC experts will judge the quality of hand hygiene in these videos, which will be adopted as ground truth in image processing. The percentage of fluorescent gel residual on hands shown in the hand scanner will be used as an objective assessment for efficacy of hand washing in individual participants.

Post-intervention assessment

The participants will take the second hand washing attempt by putting fluorescent powder on both of their hands again and then perform hand wash with videos recorded. After washing hands, participants will scan fluorescent powder remained on their hands again in a hand scanner. Participants will also be asked to fill in a questionnaire on knowledge and practice of hand hygiene as part of post-intervention assessment.

For the training purpose, after the completion of post-intervention measurements, the participants of the control group will watch the training video and repeated hand washing and scanning for the third time if they agree. But the results of their third hand washing attempt will not be included into data analysis in this study.

Randomization, allocation concealment, and blinding

Participants will be randomly assigned to the intervention groups or control group through a process of randomization performed by a statistician who will not be involved in subject recruitment. The participants will be blinded. The RAs involved in subject recruitment and the IPC experts who judge the quality of hand hygiene will be blinded to the groupings. The RAs and student assistants involved in hand hygiene video recording at the study site will not be blinded because they will be giving instructions to the participants.

ELIGIBILITY:
Inclusion Criteria:

* all year one nursing students from the Bachelor of Nursing and Bachelor of Mental Health Nursing program in School of Nursing

Exclusion Criteria:

* students with severe eczema or other extreme hand conditions will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Practice of hand hygiene | 5 minutes after hand washing
  The percentage (from 0 to 100%, the higher scores mean a worse outcome) of fluorescent gel residual on hands shown in the hand scanner will be used as an objective assessment for efficacy of hand washing in individual participants.

SECONDARY OUTCOMES:
Knowledge of hand hygiene | 10 minutes before and 10 minutes after hand washing
  Participants will be asked to fill in the pre- and post questionnaires on knowledge and practice of hand hygiene as part of intervention assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Squina International Centre for Infection Control, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared upon request to the PI.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication.
Access Criteria: The Responsible Party will review the requests.

REFERENCES:
- [Derived] Chen J, Yang L, Mak YW, O'Donoghue M, Shi C, Tsang H, Lu S, Zou J, Qin J, Xie YJ, Lai T, Li C, Cao J, Pittet D. Hand Hygiene Education Components Among First-Year Nursing Students: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2413835. doi: 10.1001/jamanetworkopen.2024.13835. PMID 38869902

DOCUMENTS (1):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT05872581/Prot_000.pdf